CLINICAL TRIAL: NCT02292186
Title: A Phase 2, Open-label Extension Study to Evaluate the Long-Term Safety, Clinical Activity, and Pharmacokinetics of ALN-TTRSC in Patients With Transthyretin (TTR) Cardiac Amyloidosis Who Have Previously Received ALN-TTRSC
Brief Title: A Extension Study to Evaluate Revusiran (ALN-TTRSC) in Patients With Transthyretin (TTR) Cardiac Amyloidosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alnylam Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALN-TTRSC-003
Record Dates: First submitted 2014-11-10; First posted 2014-11-17 (Estimated); Results first posted 2018-06-15 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-07

CONDITIONS: TTR-mediated Amyloidosis
Keywords: Cardiomyopathy; Heart Failure; FAC; Amyloid; Transthyretin; TTR; RNAi therapeutic
MeSH Terms: conditions — Cardiomyopathies; Heart Failure; Alzheimer Disease | interventions — revusiran

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Revusiran (ALN-TTRSC) (Experimental)
  Interventions: Drug: Revusiran (ALN-TTRSC)

INTERVENTIONS:
Drug: Revusiran (ALN-TTRSC)

SUMMARY:
The purpose of this study was to evaluate the safety and clinical activity of long-term dosing with revusiran (ALN-TTRSC). Dosing has been discontinued; patients are being followed-up for safety.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who previously received and tolerated revusiran (ALN-TTRSC) in the ALN-TTRSC-002 study
* Adequate liver function
* Not Pregnant or nursing

Exclusion Criteria:

* Inadequate renal function
* Uncontrolled hypertension, ischemic heart disease or clinically significant cardiac arrhythmia
* Untreated hypo- or hyperthyroidism
* Prior major organ transplant

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2014-10; Primary Completion 2017-02-22 (Actual); Study Completion 2017-02-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jared Gollob, MD, Study Director — Alnylam Pharmaceuticals
Locations (5):
- United States (3):
  - Clinical Trial Site, Boston, Massachusetts
  - Clinical Trial Site, New York, New York
  - Clinical Trial Site, Cleveland, Ohio
- Clinical Trial Site, Calgary, Alberta, Canada
- Clinical Trial Site, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Revusiran (ALN-TTRSC): All patients who received at least 1 dose of revusiran
Period: Overall Study
Arm/Group | Revusiran (ALN-TTRSC)
Started | 25
Completed | 7
Not Completed | 18

BASELINE CHARACTERISTICS:
Population: All patients who received at least 1 dose of revusiran
Arm/Group | Revusiran (ALN-TTRSC)
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.8 (6.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 21
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability Results of Long-term Dosing With ALN-TTRSC (Revusiran) Transthyretin (TTR) Cardiac Amyloidosis Patients.
Description: The proportion of subjects experiencing adverse events (AEs), serious adverse events (SAEs) and study [drug] discontinuation.
Time Frame: Day 0 up to 90 days post modified early termination visit (end of study); Mean duration of collection was 16 months
Measure: Count of Participants; unit: Participants
Arm/Group | Revusiran (ALN-TTRSC)
Number analyzed (Participants) | 25
Participants
  At least 1 AE (adverse event) | 25
  At least 1 SAE (serious adverse event) | 22
  Study discontinuation for any reason | 18

2. Primary Outcome: Serum TTR Levels
Description: Pharmacodynamic (PD) effect of long-term dosing of ALN-TTRSC on serum levels of TTR
Time Frame: Day 0 up to 90 days post modified early termination visit (end of study); Mean duration of collection was 16 months
Population: Long term samples not collected due to study termination; no data to analyze
Arm/Group | Revusiran (ALN-TTRSC)
Number analyzed (Participants) | 0

3. Secondary Outcome: Mortality
Description: Total number of deaths in the study and total number of deaths adjudicated as being related to cardiovascular causes. Deaths were adjudicated by an independent adjudication committee as cardiovascular (CV) or non-CV events.
Time Frame: Day 0 up to 90 days post modified early termination visit (end of study); Mean duration of collection was 16 months
Measure: Count of Participants; unit: Participants
Arm/Group | Revusiran (ALN-TTRSC)
Number analyzed (Participants) | 25
Participants
  Total deaths | 8
  Total CV mortality events | 6

4. Secondary Outcome: Clinical Effects of Long-term Dosing of ALN-TTRSC on Hospitalization
Description: Hospitalization events were adjudicated by an independent committee as cardiovascular (CV) or non-CV events
Time Frame: Day 0 up to 90 days post modified early termination visit (end of study); Mean duration of collection was 16 months
Measure: Count of Participants; unit: Participants
Arm/Group | Revusiran (ALN-TTRSC)
Number analyzed (Participants) | 25
Participants
  At least 1 hospitalization event on study | 17
  At least 1 CV hospitalization event | 15

5. Secondary Outcome: 6-minute Walk Test Performance
Description: Distance in meters walked in 6 minutes
Time Frame: Baseline, Month 6, and Month 12
Population: Number of participants analyzed differs from baseline to 6 and 12 months due to study discontinuations
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Revusiran (ALN-TTRSC)
Number analyzed (Participants) | 25
meters
  Change from baseline at Month 6: number analyzed (Participants) | 19
  Change from baseline at Month 6 | -20.6 (46.1)
  Change from baseline at Month 12: number analyzed (Participants) | 15
  Change from baseline at Month 12 | -104.6 (88.6)

ADVERSE EVENTS:
Time Frame: All AEs that occurred after the start of study drug administration on Day 0 (Baseline) up to 90 days post modified early termination visit (End of Study); Mean duration of collection was 16 months.
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study
Arm/Group | Revusiran (ALN-TTRSC)
All-Cause Mortality (participants affected / at risk) | 8/25
Serious Adverse Events (participants affected / at risk) | 22/25
Other Adverse Events (participants affected / at risk) | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Revusiran (ALN-TTRSC) (N=25)
Neuropathy peripheral (Nervous system disorders) | 7 (8)
Cardiac failure (Cardiac disorders) | 6 (6)
Hypotension (Vascular disorders) | 6 (6)
Blood lactic acid increased (Investigations) | 3 (3)
Cardiac failure congestive (Cardiac disorders) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pneumonia (Infections and infestations) | 3 (4)
Renal impairment (Renal and urinary disorders) | 3 (3)
Atrial fibrillation (Cardiac disorders) | 2 (2)
Cardiac arrest (Cardiac disorders) | 2 (2)
Cardiac failure acute (Cardiac disorders) | 2 (2)
Cardiogenic shock (Cardiac disorders) | 2 (2)
Cerebrovascular accident (Nervous system disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2)
Fluid overload (Metabolism and nutrition disorders) | 2 (2)
Lower respiratory tract infection (Infections and infestations) | 2 (2)
Neuralgia (Nervous system disorders) | 2 (2)
Renal failure acute (Renal and urinary disorders) | 2 (2)
Sepsis (Infections and infestations) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Lactic acidosis (Metabolism and nutrition disorders) | 1 (1)
Generalised oedema (General disorders) | 1 (3)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)
Amyloidosis (Immune system disorders) | 1 (1)
Obstructive uropathy (Renal and urinary disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Left ventricular dysfunction (Cardiac disorders) | 1 (1)
Atrial flutter (Cardiac disorders) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Large intestinal ulcer (Gastrointestinal disorders) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Myopathy (Musculoskeletal and connective tissue disorders) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Vasoplegia syndrome (Injury, poisoning and procedural complications) | 1 (1)
Completed suicide (Psychiatric disorders) | 1 (1)
Electrocardiogram QRS complex prolonged (Investigations) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Right ventricular failure (Cardiac disorders) | 1 (1)
Renal failure chronic (Renal and urinary disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Asthenia (General disorders) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Revusiran (ALN-TTRSC) (N=25)
Cough (Respiratory, thoracic and mediastinal disorders) | 12 (17)
Dizziness (Nervous system disorders) | 10 (14)
Neuropathy peripheral (Nervous system disorders) | 9 (12)
Fall (Injury, poisoning and procedural complications) | 10 (11)
Hypotension (Vascular disorders) | 4 (5)
Constipation (Gastrointestinal disorders) | 9 (10)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 (10)
Oedema peripheral (General disorders) | 9 (13)
Fatigue (General disorders) | 8 (8)
Injection site erythema (General disorders) | 8 (41)
Atrial fibrillation (Cardiac disorders) | 7 (7)
Urinary tract infection (Infections and infestations) | 7 (8)
Weight decreased (Investigations) | 7 (9)
Diarrhoea (Gastrointestinal disorders) | 6 (6)
Injection site pruritus (General disorders) | 6 (29)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 6 (7)
Blood lactic acid increased (Investigations) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 4 (4)
Fluid overload (Metabolism and nutrition disorders) | 3 (3)
Injection site pain (General disorders) | 5 (14)
International normalized ratio increased (Investigations) | 5 (8)
Nausea (Gastrointestinal disorders) | 5 (5)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5 (7)
Renal failure acute (Renal and urinary disorders) | 4 (5)
Lower respiratory tract infection (Infections and infestations) | 3 (5)
Contusion (Injury, poisoning and procedural complications) | 4 (4)
Injection site swelling (General disorders) | 4 (16)
Liver function test abnormal (Investigations) | 4 (4)
Orthostatic hypotension (Vascular disorders) | 4 (6)
Pneumonia (Infections and infestations) | 2 (2)
Vitamin A decreased (Investigations) | 4 (4)
Cardiac failure (Cardiac disorders) | 4 (4)
Gamma-glutamyltransferase increased (Investigations) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 2 (3)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Blood creatinine increased (Investigations) | 2 (2)
Blood urea increased (Investigations) | 2 (2)
Sinusitis (Infections and infestations) | 2 (2)
Urinary retention (Renal and urinary disorders) | 2 (2)
Excoriation (Injury, poisoning and procedural complications) | 2 (2)
Tooth infection (Infections and infestations) | 2 (2)
Flushing (Vascular disorders) | 2 (8)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (4)
Rash (Skin and subcutaneous tissue disorders) | 2 (4)
Laceration (Injury, poisoning and procedural complications) | 2 (2)
Joint swelling (Musculoskeletal and connective tissue disorders) | 3 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Injection site discoloration (General disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Bronchitis (Infections and infestations) | 3 (3)
Abdominal discomfort (Gastrointestinal disorders) | 3 (3)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (2)
Pericardial effusion (Cardiac disorders) | 2 (2)
Depression (Psychiatric disorders) | 3 (3)
Rales (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Pyrexia (General disorders) | 2 (2)
Injection site inflammation (General disorders) | 2 (3)
Gout (Metabolism and nutrition disorders) | 2 (2)
Increased tendency to bruise (Skin and subcutaneous tissue disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (3)
Onychomycosis (Infections and infestations) | 2 (2)
Carpal tunnel syndrome (Musculoskeletal and connective tissue disorders) | 2 (2)
Erectile dysfunction (Reproductive system and breast disorders) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3)
Headache (Nervous system disorders) | 3 (3)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Tremor (Nervous system disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 2 (2)
Dysgeusia (Nervous system disorders) | 2 (2)
Traumatic haematoma (Injury, poisoning and procedural complications) | 2 (2)
Vertigo (Ear and labyrinth disorders) | 2 (2)
Intervertebral disk degeneration (Musculoskeletal and connective tissue disorders) | 2 (2)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 (2)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 2 (2)
Injection site haematoma (General disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
Safety and efficacy data are difficult to interpret due to the limited numbers of patients completing the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2016-03-25): https://cdn.clinicaltrials.gov/large-docs/86/NCT02292186/Prot_000.pdf
  • Statistical Analysis Plan (2014-10-23): https://cdn.clinicaltrials.gov/large-docs/86/NCT02292186/SAP_001.pdf